CLINICAL TRIAL: NCT03380091
Title: Metformin, Vitamin D, and Depression in Polycystic Ovary Syndrome (PCOS) Trial: The MINDD Trial
Brief Title: Metformin, Vitamin D, and Depression in Polycystic Ovary Syndrome (PCOS) Trial
Acronym: MINDD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-22550
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: PCOS; Depression; Vitamin D Deficiency; Insulin Resistance
Keywords: PCOS; Depression; Vitamin D; Insulin Resistance; Anxiety; Quality of life; Mood disorders
MeSH Terms: conditions — Depression; Vitamin D Deficiency; Insulin Resistance; Anxiety Disorders; Mood Disorders | interventions — Metformin; Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Metformin 1000 mg PO bid
  Interventions: Drug: Metformin
- Vitamin D (Cholecalciferol) (Experimental): Cholecalciferol 5,000 IU PO daily
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Metformin — Oral medication daily
  Other Names: Glucophage; Glucophage XR; Fortamet; Glumetza
  Arms: Metformin
Drug: Vitamin D — Oral medication daily
  Other Names: Cholecalciferol
  Arms: Vitamin D (Cholecalciferol)

SUMMARY:
Open-label randomized clinical trial assessing the efficacy of Metformin versus Vitamin D in improving symptoms of depressed mood in polycystic ovary syndrome.

DETAILED DESCRIPTION:
This is a single center, open-label, randomized, pilot clinical trial. Women with polycystic ovary syndrome and depressed mood, who are insulin resistant and vitamin D insufficient are eligible. Subjects are randomly assigned to one of two interventions: Vitamin D versus metformin. Subjects are followed with questionnaires and a final wrap-up clinic visit with a physician. The study duration is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic Ovary Syndrome diagnosis (Rotterdam Criteria)
* Vitamin D insufficiency (serum Vitamin D <30 ng/mL)
* Insulin resistance
* Mild or greater severity of depression by Beck Depression Inventory-II

Exclusion Criteria:

* Current metformin use
* Vitamin D supplementation of > 50,000 IU following confirmation of Vitamin D insufficiency
* Insulin-dependent diabetes mellitus
* Pregnancy or breastfeeding
* Untreated hypothyroidism
* Current active substance abuse
* Other major medical comorbidity: renal or hepatic dysfunction, severe pulmonary
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 5 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 5 participants that were enrolled in the trial, all were randomized and assigned to treatment arms. 3 were assigned to the Vitamin D supplement arm and 2 were assigned to the Metformin arm.
Period: Overall Study
Arm/Group | Vitamin D (Cholecalciferol) | Metformin
Started | 3 | 2
Began Arm Treatment | 1 (1 participant withdrew after completing baseline measures and another withdrew just after enrolling.) | 1 (1 of the 2 participant assigned to Metformin withdrew from the study just after enrolling.)
Completed | 1 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Although 3 participants were assigned to Vitamin D, one dropped out just after enrollment and arm assigment and another dropped out after completing baseline time point measures, thus only one participant in the Vitamin D arm had data available for outcome measures analysis. Although 2 participants were assigned to Metformin, one dropped out just after enrollment and arm assignment, thus only one participant in the Metformin arm had data available for outcome measures analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D (Cholecalciferol) | Metformin | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Fasting Insulin [Mean (Standard Deviation); unit: μIU/mL] — Fasting blood insulin levels were assayed by Quest Diagnostics. Time point: Baseline, pre-intervention
  Optimal Reference range:
  Fasting 2.0-19.6 μIU/mL
  μIU/mL | 14.2 (4.6) | 32 (0) | 20.13 (9.19)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] — Fasting blood glucose levels were assayed by Quest Diagnostics. Time point: Baseline, pre-intervention
  Optimal Reference range:
  Fasting 65-99 mg/dL
  mg/dL | 90.5 (3.5) | 83 (0) | 88 (4.54)
Fasting Insulin Resistance [Mean (Standard Deviation); unit: units on a scale] — Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) will be used to calculate Insulin Resistance based on fasting glucose (mg/dL) and fasting insulin (μIU/mL) blood serum assays tested at Quest Diagnositcs.
  Time point: Baseline, pre-intervention HOMA-IR = Fasting Insulin (uIU/mL) x Fasting Glucose (mg/dL). Healthy range is between 0.5-1.4. Values below 1.0 indicate insulin sensitivity and are optimal. Values greater than 1.9 indicate clinically significant insulin resistance.
  units on a scale | 3.12 (0.92) | 6.6 (0) | 4.28 (1.80)
Vitamin D, 25 hydroxy [Mean (Standard Deviation); unit: ng/mL] — Vitamin D, 25-hydroxy blood serum assays will be tested at Quest Diagnostics. Time period: baseline, pre-intervention
  Reference ranges:
  optimal 30-100 ng/mL Insufficient 20-29 ng/mL deficient <20ng/mL
  ng/mL | 21.5 (2.5) | 21 (0) | 21.33 (2.05)
Beck Depression Inventory (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — BDI-II is a validated self-reported instrument of 21 questions which are each scored 0-3. Total scores range from 0-63, with higher score totals indicating more severe depression symptoms.
  Time period: baseline; pre-intervention
  Score ranges:
  {0-9: indicates minimal depression; 0-18: indicates mild depression; 19-29: indicates moderate depression; 30-63: indicates severe depression}.
  units on a scale | 21.5 (4.5) | 18 (0) | 20.33 (4.02)
State-Trait Anxiety Inventory Score (STAI-S) [Mean (Standard Deviation); unit: units on a scale] — STAI-S is a validated self-reported instrument of 20 questions. Time period: baseline, pre-intervention
  Range of scores for the State Anxiety (STAI-S) subtest is 20-80, the higher score indicating greater anxiety. A threshold point score of 39-40 has been suggested by recent literature to detect clinically significant symptoms
  units on a scale | 54.5 (3.5) | 44 (0) | 51 (5.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depression Score on the Beck Depression Inventory (BDI-II) at 12 Weeks
Description: BDI-II is a validated self-reported instrument of 21 questions which are each scored 0-3. Total scores range from 0-63, with higher score totals indicating more severe depression symptoms. {0-9: indicates minimal depression; 0-18: indicates mild depression; 19-29: indicates moderate depression; 30-63: indicates severe depression}. Change = Week 12 total score - Baseline week score
Time Frame: Baseline & 12 weeks
Population: In both the Vitamin D and the Metformin arms, only 1 participant in each arm was analyzed for Change in Depression from Baseline as only 1 participant in each arm participated through to week 12. A Change could not be calculated for the other 3 participants as no week 12 scores were available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D (Cholecalciferol) | Metformin
Number analyzed (Participants) | 1 | 1
score on a scale | -8 (0) | 7 (0)

2. Secondary Outcome: Changes From Baseline Week in Insulin Resistance Score at Week 12.
Description: Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) will be used to calculate Insulin Resistance based on fasting glucose (mg/dL) and fasting insulin (μIU/mL) blood serum assays tested at Quest Diagnostics. HOMA-IR = Fasting Insulin (uIU/mL) x Fasting Glucose (mg/dL). Healthy range is between 0.5-1.4. Values below 1.0 indicate insulin sensitivity and are optimal. Values greater than 1.9 indicate clinically significant insulin resistance.
Time Frame: Baseline week & week 12
Population: In both the Vitamin D and the Metformin arms, only 1 participant in each arm was analyzed for Change in Insulin Resistance from Baseline as only 1 participant in each arm participated through to week 12. A Change could not be calculated for the other 3 participants as no week 12 serum insulin and glucose test results were available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vitamin D (Cholecalciferol) | Metformin
Number analyzed (Participants) | 1 | 1
units on a scale | 0.81 (0) | -1.2 (0)

3. Secondary Outcome: Change From Baseline in State-Trait Anxiety Inventory Score (STAI-S) at 12 Weeks
Description: STAI-S is a validated self-reported instrument of 20 questions. Range of scores for the State Anxiety (STAI-S) subtest is 20-80, the higher score indicating greater anxiety. A threshold point score of 39-40 has been suggested by recent literature to detect clinically significant symptoms. Change = Week 12 total score - Baseline week score
Time Frame: Baseline week & Week 12
Population: In both the Vitamin D and the Metformin arms, only 1 participant in each arm was analyzed for a Change in Anxiety scores from Baseline as only 1 participant in each arm participated through to week 12. A Change could not be calculated for the other 3 participants as no week 12 scores were available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metformin | Vitamin D (Cholecalciferol)
Number analyzed (Participants) | 1 | 1
score on a scale | 0 (0) | 10 (0)

4. Secondary Outcome: Changes From Baseline Week in Vitamin D 25-hydroxy Levels at Week 12.
Description: Vitamin D, 25-hydroxy blood serum assays will be tested at Quest Diagnostics. Changes in values from baseline week to week 12 will be calculated.
  Reference ranges:
  optimal 30-100 ng/mL Insufficient 20-29 ng/mL deficient <20ng/mL
Time Frame: Baseline week & week 12
Population: In both the Vitamin D and the Metformin arms, only 1 participant in each arm was analyzed for Change in Vitamin D serum levels from Baseline as only 1 participant in each arm participated through to week 12. A Change could not be calculated for the other 3 participants as no week 12 serum Vitamin D test results were available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D (Cholecalciferol) | Metformin
Number analyzed (Participants) | 1 | 1
mg/dL | 11 (0) | -5 (0)

ADVERSE EVENTS:
Time Frame: Study activity participation window of 12 weeks.
Description: AE and SAE definition meet clinicaltrials.gov definitions
  Investigators will carefully track serious adverse events and all of these events will be reported to the DSM at scheduled meetings. Grade 4 adverse events will be reported to the DSM within 24 hours of receipt by the Study Coordinator. Adverse events meeting IRB reporting criteria (adverse event that are definitely, probably, or possibly related to the research AND serious OR unexpected) will be reported within 5 working days.
Arm/Group | Vitamin D (Cholecalciferol) | Metformin
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
Feasibility of recruitment and participant completion determined to be too low to continue the study and the trial was terminated early, resulting in only 2 of the 5 enrolled participants completing the trial. This lead to only two subjects will full data and one subject with partial data being analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT03380091/Prot_SAP_000.pdf